CLINICAL TRIAL: NCT04718220
Title: Safety, Testing/Transmission, and Outcomes in Pregnancies With COVID-19
Acronym: STOPCOVID19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Mercy Research (Other)
Responsible Party: Principal Investigator, Jeannie Kelly, Assistant Professor, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202012075
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Covid19; Pregnancy Related; Maternal Complication of Pregnancy; Coronavirus; Neonatal Infection; Prenatal Stress; Preterm Birth
Keywords: pregnancy; COVID-19; SARS-CoV-2; antibody testing; pregnancy complication; maternal complication; neonatal complication; mother-to-fetal transmission; placental pathology; prenatal; stress; SARS-CoV-2 testing; social determinants of health
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Premature Birth; Pregnancy Complications | interventions — Antibody Formation

STUDY DESIGN:
Intervention Model Description: This is a prospective study that will enroll two cohorts of pregnant women: 1) exposed (SARS-CoV-2 positive), and 2) unexposed (SARS-CoV-2 negative as defined by antibody testing at the beginning of pregnancy, every trimester, and at delivery). Women who initially enroll as unexposed but later test positive for SARS-CoV-2 antibodies will cross over to the exposed cohort. Outcomes will be compared between the two cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unexposed (SARS-CoV-2 negative) cohort (Placebo Comparator): Women who do not experience laboratory-confirmed SARS-CoV-2 infection during pregnancy.
  Interventions: Diagnostic Test: Antibody testing for SARS-CoV-2 IgG
- Exposed (SARS-CoV-2 positive) cohort (Active Comparator): Women who experience laboratory-confirmed SARS-CoV-2 infection during pregnancy.
  Interventions: Diagnostic Test: Testing for SARS-CoV-2 RNA; Diagnostic Test: Testing for SARS-CoV-2 IgM/IgG

INTERVENTIONS:
Diagnostic Test: Antibody testing for SARS-CoV-2 IgG — Women enrolled into the unexposed (SARS-CoV-2 negative) cohort will undergo testing for SARS-CoV-2 IgG antibodies at enrollment, every trimester of pregnancy, and during delivery hospitalization.
  Arms: Unexposed (SARS-CoV-2 negative) cohort
Diagnostic Test: Testing for SARS-CoV-2 RNA — Women in the exposed (SARS-CoV-2 positive) cohort will undergo testing of placental tissue, umbilical cord blood, amniotic tissue, and neonates for SARS-CoV-2 RNA, as available.
  Arms: Exposed (SARS-CoV-2 positive) cohort
Diagnostic Test: Testing for SARS-CoV-2 IgM/IgG — Women in the exposed (SARS-CoV-2 positive) cohort will undergo testing of umbilical cord blood for SARS-CoV-2 IgG and IgM antibodies, as available.
  Arms: Exposed (SARS-CoV-2 positive) cohort

SUMMARY:
Pregnant women are a vulnerable and high-risk population, as COVID-19 is associated with an increased risk preterm birth, cesarean section, and maternal critical care. This study will examine the factors that impede testing for SARS-CoV-2 (the causative virus among pregnant women), help determine optimal testing strategies by evaluating the necessity of testing for asymptomatic disease in pregnancy, inform prenatal care plans by assessing the full impact of infection, and contribute to a provider's ability to counsel women and create prenatal care plans if they are pregnant or considering pregnancy.

DETAILED DESCRIPTION:
Pregnant women are a vulnerable and high-risk population, as COVID-19 is associated with an increased risk of preterm birth, cesarean section, and maternal intensive care. The objectives of this study are to: (a) evaluate the full impact of SARS-CoV-2 in pregnancy to inform testing strategies, (b) examine the factors that impede testing during pregnancy, and (c) use study data to devise implementation strategies that improve SARS-CoV-2 testing in pregnancy and prenatal care during the pandemic. Investigators will prospectively enroll two cohorts of pregnant women: 1) exposed (SARS-CoV-2 positive), and 2) unexposed (SARS-CoV-2 negative as defined by antibody testing at the beginning of pregnancy, every trimester, and at delivery). Women who initially enroll as unexposed but later test positive for SARS-CoV-2 antibodies will cross over to the exposed cohort. In Aim 1, investigators will evaluate patients' and providers' perceptions of SARS-CoV-2 testing during pregnancy and the influence of COVID-19 on maternal care-seeking behavior and anxiety via surveys and semi-structured interviews. In Aim 2, investigators will determine the effect of SARS-CoV-2 infection during pregnancy on the risk of preterm birth and other adverse pregnancy outcomes in symptomatic and asymptomatic disease. It is hypothesized that SARS-CoV-2 infection will increase the risk of preterm birth by 12%. In Aim 3, investigators will estimate the risk of mother-to-fetus SARS-CoV-2 transmission and viral presence in umbilical cord blood, placenta, and amniotic fluid by assaying for viral RNA in the neonate, cord blood, and placenta. Collectively, Aims 1-3 will be interpreted by investigators, the Scientific Advisory Board and the Community Advisory Board who will apply data to devising targeted implementation strategies designed for rapid community dissemination to improve testing and prenatal care.

ELIGIBILITY:
Inclusion Criteria for exposed (SARS-CoV-2 positive) cohort:

* Viable intrauterine pregnancy
* Seroconversion or SARS-CoV-2 IgG antibodies or positive RT-PCR for SARS-CoV-2 during current pregnancy

Exclusion Criteria for exposed (SARS-CoV-2 positive) cohort:

* No viable intrauterine pregnancy
* No history of SARS-CoV-2 infection during pregnancy

Inclusion Criteria for unexposed (SARS-CoV-2 negative) cohort:

* Viable intrauterine pregnancy
* No history of SARS-CoV-2 infection prior to pregnancy

Exclusion Criteria for unexposed (SARS-CoV-2 negative) cohort:

* No viable intrauterine pregnancy
* Detection of SARS-CoV-2 IgG antibodies at enrollment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of preterm delivery | 20 weeks gestation until childbirth
  Childbirth prior to 37 weeks of pregnancy, to be determined in accordance to standard pregnancy dating and the established estimated due date.

SECONDARY OUTCOMES:
Rate of preeclampsia | After 20 weeks gestation and up to 6 weeks postpartum
  Standard definitions will be used (new-onset presence of elevated blood pressure > 140 systolic or > 90 diastolic separated by >4 hours and new onset proteinuria after 20 weeks of pregnancy or evidence of severe features of preeclampsia).
Rate of gestational hypertension | After 20 weeks gestation and up to 6 weeks postpartum
  Standard definitions of gestational hypertension will be used (new-onset presence of elevated blood pressure > 140 systolic or > 90 diastolic separated by >4 hours without proteinuria after 20 weeks of pregnancy).
Rate of cesarean section | Time of delivery
  Delivery via a cesarean section operation.
Rate of stillbirth | Between 20 weeks gestation and childbirth
  Fetal demise in utero after 20 weeks gestation.
Rate of fetal growth restriction | Between conception and childbirth
  Estimated fetal weight by sonographic assessment less than the 10th percentile for gestational age.
Rate of fetal hydrops | Between conception and childbirth
  The presence of abnormally located fluid collections in two or more areas in the fetal body (i.e., fetal ascites and pericardial effusion) or one abnormal fluid collection plus fetal skin thickening.
Rate of oligohydramnios | Between conception and childbirth
  Estimated amniotic fluid index less than 5 or estimated deepest vertical pocket (no presence of umbilical cord) less than 2 by sonographic assessment.
Perinatal death | During the pregnancy after 20 weeks of pregnancy to 21 days after delivery
  Fetal or neonatal death occurring after 20 weeks gestation and up to 21 days of life.
Rate of premature preterm rupture of membranes | Between conception and 36 weeks 6 days of pregnancy
  Rupture of membranes prior to 37 weeks gestation.
Rate of neonatal intensive care unit (NICU) admission | After delivery of newborn during delivery hospitalization
  Admission of the newborn to the NICU after delivery during delivery hospitalization.
Rate of neonatal sepsis | After delivery of newborn during delivery hospitalization up to 6 weeks of life
  Clinical syndrome that includes systemic signs of infection and bacteremia.
Rate of oxygen therapy | After delivery of newborn during delivery hospitalization up to 6 weeks of life
  Use of oxygen therapy for the newborn after delivery during delivery hospitalization.
Percentage of infants with low 5-minute Apgar | At time of delivery
  Five minute Apgar less than 7. Maximum 10, minimum 0. Higher scores typically have improved outcomes.
Percentage of infants with abnormal umbilical cord gas | At time of delivery
  pH of arterial blood of umbilical cord blood less than 7 and/or base excess greater than -12.
Low birth weight | At time of delivery
  Weight at birth less than 2,500 grams.
Confirmed congenital infection | Testing will be conducted at time of delivery.
  SARS-CoV-2 RNA detection in the umbilical cord blood, in amniotic fluid if collected before rupture of membranes or in neonatal nasopharyngeal swabs collected both immediately after birth (and after cleaning of the infant).
Probable congenital infection | At time of delivery
  SARS-CoV-2 RNA detection in the neonatal nasopharyngeal swabs collected immediately after birth (after cleaning of infant) and in the fetal side of the placenta.
Possible congenital infection | At time of delivery
  Anti-SARS-CoV-2 IgM antibodies detection in the umbilical cord blood but no SARS-CoV-2 RNA detected in the neonate.

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Foeller, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Medical Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No